CLINICAL TRIAL: NCT00413114
Title: A Phase II Study of Obatoclax Mesylate (GX15-070MS) in Patients With Previously-Untreated Myelodysplastic Syndromes (MDS) With Anemia and/or Thrombocytopenia
Brief Title: Safety and Efficacy of Obatoclax Mesylate (GX15-070MS)for the Treatment of Myelodysplastic Syndromes (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gemin X (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM013
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — obatoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obatoclax Mesylate (Experimental): Obatoclax Mesylate 30mg
  Interventions: Drug: Obatoclax mesylate (GX15-070MS)

INTERVENTIONS:
Drug: Obatoclax mesylate (GX15-070MS)

SUMMARY:
Defects in the apoptotic process can lead to the onset of cancer by allowing cells to grow unchecked when an oncogeneic signal is present. Obatoclax is designed to restore apoptosis through inhibition of the Bcl-2 family of proteins, thereby reinstating the natural process of cell death that is often inhibited in cancer cells.

This is a multi-center, open-label, Phase II study of obatoclax administered in 2-week cycles to patients with previously-untreated Myelodysplastic Syndromes with anemia and/or thrombocytopenia. Treatment may be administered on an outpatient basis. No investigational or commercial agents or therapies other than those described herein may be administered with the intent to treat the patient's malignancy. Supportive care measures including those directed at controlling symptoms resulting from Myelodysplastic Syndromes are allowed

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation of Myelodysplastic Syndromes (MDS)
* Patients must have had no prior systemic therapy
* Must have normal organ functions
* Must have the ability to understand and willingness to sign a written informed consent form

Exclusion Criteria:

* Must not be a result of prior chemotherapy and/or radiotherapy for another malignancy
* No other agents or therapies administered in the intent to treat
* Uncontrolled, intercurrent illness
* Pregnant women and women who are breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-12; Primary Completion 2009-02 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
International Working Group (IWG) Response Criteria for MDS | 52 weeks
  Determine the response rate according to bone marrow blast count less than or equal to 10%

SECONDARY OUTCOMES:
Peripheral blood counts; Bone marrow aspirates and biopsies; Transfusions and growth factor requirements | 52 weeks
  hemoglobin level less than 10 g/dL and or platelets less than 50 x 10 9/L. Eastern Cooperative Onocology Group (ECOG) performance status: 0 fully active-2 ambulatory 50% of the time; and total bilirubin less than or equal to 2 mg/dL; normal limits of SGOT/SGPT and creatinine according to laboratory standards

CONTACTS AND LOCATIONS:
Overall Officials: Mark Berger, MD, Study Director — Gemin X, Inc.
Locations (22):
- United States (17):
  - Stanford University, Stanford, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - James A. Haley Veterans Hospital, Tampa, Florida
  - Emory University School of Medicine/ Winship Cancer Center, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Michigan State University, Breslin Cancer Center CTO, Lansing, Michigan
  - Hematology-Oncology Centers of the Northern Rockies, Billings, Montana
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - Pacific Oncology, Portland, Oregon
  - The West Clinic, Memphis, Tennessee
  - Sarah Cannon Cancer Research Institute, Nashville, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - Texax Oncology, P.A., Presbyterian/ Mary Crowley Clinical Research Centers, Dallas, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
  - MD Anderson Cancer Center (Protocol 2006-0688), Houston, Texas
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - QEII HSC, Halifax, Nova Scotia
  - Princess Margaret Hospital, Toronto, Ontario
  - Hospital Notre-Dame du Chum, Montreal, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Arellano ML, Borthakur G, Berger M, Luer J, Raza A. A phase II, multicenter, open-label study of obatoclax mesylate in patients with previously untreated myelodysplastic syndromes with anemia or thrombocytopenia. Clin Lymphoma Myeloma Leuk. 2014 Dec;14(6):534-9. doi: 10.1016/j.clml.2014.04.007. Epub 2014 Jun 12. PMID 25052051